CLINICAL TRIAL: NCT00606853
Title: Enhanced and Attendance-based Prize CM in Community Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 04-008; P50DA009241 (NIH)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Cocaine Dependence
Keywords: Substance abuse; Contingency Management
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Standard Treatment plus prize contingency management for abstinence with an expected probability of winning about $250 in prizes and twice-weekly breath and urine samples.
  Interventions: Behavioral: Contingency Management
- 2 (Experimental): Standard Treatment plus prize contingency management for abstinence with an expected probability of winning about $560 in prizes and twice-weekly breath and urine samples.
  Interventions: Behavioral: Contingency Management
- 3 (Experimental): Standard Treatment plus prize contingency management for attendance with an expected probability of winning about $250 in prizes and twice-weekly breath and urine samples.
  Interventions: Behavioral: Contingency Management
- 4 (No Intervention): Standard Treatment

INTERVENTIONS:
Behavioral: Contingency Management — Rewards valued $1-$100 for abstinence or treatment attendance
  Arms: 1; 2; 3

SUMMARY:
The purpose of this study is to address the conditions under which prize contingency management (CM) for abstinence and attendance may improve outcomes of cocaine-dependent patients.

For patients who initiate treatment with a cocaine-positive urine specimen, we will evaluate the efficacy of two CM procedures relative to standard, non-CM treatment. The two CM procedures will be provided as additions to standard care and will reinforce drug abstinence but will differ in expected magnitudes of prizes patients can earn, especially during early stages of abstinence. They will provide expected magnitudes of winning about $250 and $560, respectively. We expect that both CM conditions will improve retention and abstinence relative to the standard treatment, non-CM condition. If the enhanced CM condition engenders better outcomes than the $250 CM condition, this finding would suggest that patients initiating treatment while actively using cocaine may best be treated with relatively high reinforcement prize CM as an adjunct to standard care.

For patients who initiate treatment with a cocaine-negative urine specimen, we will evaluate the efficacy of a CM procedure that reinforces treatment attendance. The expected magnitude of winnings will be about $250, and again CM treatment will be in addition to standard care. This CM condition will be compared to standard treatment without CM as well as to a CM treatment that provides a similar magnitude of reinforcement, but contingent upon abstinence. Results from this study will inform an important clinical question of whether simply reinforcing attendance can improve clinical outcomes. Increased retention may result in greater exposure to therapeutic processes that may reduce drug use, especially among patients who begin treatment having already achieved some abstinence. We will also evaluate the cost-effectiveness of CM by examining the effects of the interventions on hospitalizations, medical and psychiatric care, criminal justice costs, and productivity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Current DSM-IV diagnosis of cocaine dependence
* A cocaine-positive urine sample submitted during the first two scheduled treatment days at the center
* Willing to provide names, addresses and phone numbers of individuals to assist in locating the patient for follow-up evaluations
* English speaking
* Willing to sign informed consent.

Exclusion Criteria:

* Serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, bipolar disorder, severe or psychotic major depression, or suicide risk)
* Dementia (<23 on the Mini Mental State Exam; Folstein et al. 1975)
* In recovery from pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2003-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
longest continuous period of cocaine abstinence | baseline and at each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health Center
Locations (1):
- UConn Health Center, Farmington, Connecticut, United States